CLINICAL TRIAL: NCT05377242
Title: Curcumin, Resveratrol, and Stinging Nettle as Treatments for Gulf War Illness
Brief Title: Curcumin, Resveratrol, and Stinging Nettle as Treatments for GWI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jarred Younger, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: GW210009; W81XWH-22-1-0420 (Other Grant/Funding Number: GWIRP)
Record Dates: First submitted 2022-04-19; First posted 2022-05-17 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Gulf War Illness
Keywords: Gulf War Illness; Botanicals; Remote; Clinical Trial; Curcumin; Resveratrol; Stinging Nettle
MeSH Terms: interventions — Curcumin; Resveratrol; stinging nettle lectin

STUDY DESIGN:
Intervention Model Description: The study uses a prospective, pseudo-randomized, placebo-controlled, blinded, within-person clinical trial design. Individuals will be randomized in a double-blind fashion to either the curcumin, resveratrol, or stinging nettle treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, the study PI, and the main research team will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gulf War Veterans, Curcumin (Experimental): All GWI Veterans will undergo the same screening and experimental procedures. Participants must meet both the Kansas and CDC (Centers for Disease Control and Prevention) Case Definitions of GWI. Participants must have been deployed to the Persian Gulf Region during the 1990-1991 Gulf War, meet symptom domain criteria, and not have exclusionary medical conditions. This trial tests three interventions, which are all tested independently. Participants will receive only one of the three interventions. The curcumin, resveratrol, and stinging nettle trials all follow the same design and procedures.
  Participants will complete one month of baseline, eight months of capsules, and one month of endline measurements.
  Interventions: Dietary Supplement: Curcumin
- Gulf War Veterans, Resveratrol (Experimental): All GWI Veterans will undergo the same screening and experimental procedures. Participants must meet both the Kansas and CDC (Centers for Disease Control and Prevention) Case Definitions of GWI. Participants must have been deployed to the Persian Gulf Region during the 1990-1991 Gulf War, meet symptom domain criteria, and not have exclusionary medical conditions. This trial tests three interventions, which are all tested independently. Participants will receive only one of the three interventions. The curcumin, resveratrol, and stinging nettle trials all follow the same design and procedures.
  Participants will complete one month of baseline, eight months of capsules, and one month of endline measurements.
  Interventions: Dietary Supplement: Resveratrol
- Gulf War Veterans, Stinging Nettle (Experimental): All GWI Veterans will undergo the same screening and experimental procedures. Participants must meet both the Kansas and CDC (Centers for Disease Control and Prevention) Case Definitions of GWI. Participants must have been deployed to the Persian Gulf Region during the 1990-1991 Gulf War, meet symptom domain criteria, and not have exclusionary medical conditions. This trial tests three interventions, which are all tested independently. Participants will receive only one of the three interventions. The curcumin, resveratrol, and stinging nettle trials all follow the same design and procedures.
  Participants will complete one month of baseline, eight months of capsules, and one month of endline measurements.
  Interventions: Dietary Supplement: Stinging Nettle

INTERVENTIONS:
Dietary Supplement: Curcumin — Curcumin (chemical C21H20O6) is derived from turmeric (Curcuma longa) root extract, standardized to contain 95% curcuminoids. The greatest obstacle with curcumin is its poor natural bioavailability. To help circumvent that issue, a piperazine is included as black pepper 5.3mg (Piper nigrum) fruit extract standardized to 95% piperine. The botanical we are using is provided by Pure Encapsulations. Curcumin being used in this study is a commercially available dietary supplement and is classified as food by the FDA instead of a drug.
  100 participants will be randomized to receive curcumin. Participants will receive placebo, low-dose (500 mg/day), medium-dose (1000 mg/day), and/or high dose (2000 mg/day) curcumin in a randomized order.
  Arms: Gulf War Veterans, Curcumin
Dietary Supplement: Resveratrol — Resveratrol (chemical C14H12O3) is provided as 99% Pure Trans-Resveratrol (MegaResveratrol) from polygonum cuspidatum root). Resveratrol being used in this study is a commercially available dietary supplement and is classified as food by the FDA instead of a drug.
  100 participants will be randomized to receive resveratrol. Participants will receive placebo, low-dose (250 mg/day), medium-dose (500mg/day), and/or high dose (1000mg/day) resveratrol in a randomized order.
  Arms: Gulf War Veterans, Resveratrol
Dietary Supplement: Stinging Nettle — Stinging nettle is derived from nettle (Urtica spp) leaf. The botanical we are using is provided by Pure Encapsulations. Stinging Nettle being used in this study is a commercially available dietary supplement and is classified as food by the FDA instead of a drug.
  100 participants will be randomized to receive stinging nettle. Participants will receive placebo, low-dose (435mg/day), medium-dose (870mg/day), and/or high dose (2610mg/day) stinging nettle in a randomized order.
  Other Names: Urtica dioica
  Arms: Gulf War Veterans, Stinging Nettle

SUMMARY:
This project's objective is to identify effective treatments for Gulf War Illness (GWI). The project tests three potential treatments: curcumin, stinging nettle, and resveratrol. The project uses a decentralized clinical trial (DCT) design in which individuals can participate from anywhere in the United States. Recruitment efforts will be designed to obtain a geographically and demographically diverse study sample.

DETAILED DESCRIPTION:
The project is funded by the Congressionally Directed Medical Research Programs (CDMRP) of the U.S. Department of Defense.

The study uses a prospective, pseudo-randomized, placebo-controlled, blinded, within-person clinical trial design. The trials are conducted decentralized, with all protocols performed remotely. Three-hundred individuals will be recruited in the study.

Recruitment for this study will come from a database of participant who have agreed to be contacted about future studies from our previous studies. Participants will also be recruited through the Gulf War Illness Clinical Trials and Intervention Consortium (GWICTIC) through our collaboration with Nova Southeastern University. The Consortium includes a database of individuals with Gulf War Illness who had agreed to be contacted for research studies. No other information will be shared with Nova Southeastern University unless specified and agreed upon. We will also use social media advertisements in partnership with High Level Marketing to recruit for this trial.

In accordance with the Institute of Medicine (IOM) 2014 guidance, participants must meet both the Kansas and CDC (Centers for Disease Control and Prevention) Case Definitions of GWI. Participants must have been deployed to the Persian Gulf Region during the 1990-1991 Gulf War, meet symptom domain criteria, and not have other exclusionary medical conditions.

All potential participants will fill out a online screening survey to assess eligibility. If they are deemed eligible for consent, participants will undergo a zoom meeting with a member of the study staff to sign the consent form. During that meeting, the study staff will explain the consent form in detail and answer any questions about the study or the consent form. The consenting process will follow the same procedure as typically done in face-to-face consenting, and the consent form will be digitally signed during or within 24 hours after the meeting. After providing informed consent, participants will take a post-consent survey to confirm eligibility before entering the study protocol.

Participants will also be required to obtain safety tests via LabCorp or Quest Diagnostics to assess renal and hepatic function, along with collecting C-Reactive Protein readings. Because kidney and liver function are important in the metabolism and excretion of the botanicals, it must be determined that these systems can tolerate the addition of a new daily treatment. All participants will received a baseline and mid-point test of kidney and liver function. Individuals with abnormal results on these tests will not proceed with the study or receive study botanicals. Participants can obtain the tests either at a local LabCorp or Quest Diagnostics site to have blood drawn for standard hepatic and renal panels. The hepatic panel includes measuring protein, albumin, globulin, albumin/globulin ratio, total bilirubin, indirect bilirubin, alkaline phosphatase, aspartate transaminase, and alanine transaminase. Results from the blood test will be sent to the participant at their request and to the study coordinator to confirm eligibility. The information will be de-identified and only associated with the individualized study identifier.

If eligible, participants will be randomly assigned a botanical in a double-blind fashion. Participants will then begin the baseline phase of 30 days. During that time, they will complete all baseline questionnaires and will also begin the weekly symptom severity reports and primary outcome measures. A research team member will speak with the participant to set up their electronic device connections and will verify the information is received. Participants will complete all weekly measures on a computer, tablet, or phone. Individuals without an appropriate device will be sent one by the research team. The VR-12 and PGIC secondary outcomes will be given once per week during the weekly questionnaire. The 30-day period will serve as the baseline phase for all analyses. During the baseline phase and after checking that there were no exclusionary kidney or liver concerns, participants will be sent capsules. Capsules will be sent via FedEx in blister packs that indicate what order to take the botanicals. The first shipment of capsules will contain two months of capsules. On Day 31, individuals will being taking the assigned capsules in the morning and again in the evening. During this time, they will continue completing weekly symptom reports, and weekly primary and secondary outcome reports. Participants will complete one month of baseline, eight months of capsules, and one month of endline. At Day 300, their participation will be successfully completed, and they will be fully debriefed by a member of the study team soon after completion.

Consented individuals will be randomized in a double-blind fashion to either the curcumin, resveratrol, or stinging nettle treatment. The curcumin, resveratrol, and stinging nettle trials all follow the same design and procedures. Participants will be blinded not only to the botanical they receive, but also to the schedule of receiving placebo and dosage changes. The randomization schedule will be held by Dr. Nancy Klimas and Dr. Amanpreet Cheema from Nova Southeastern University.

Placebo capsules will be created to keep the same appearance to treatment capsules. Both placebo (microcrystalline cellulose) and active treatment capsules will be over-encapsulated with the same gel caps. Participants will take the same number of capsules in the morning and night throughout participation so that individuals cannot determine when active treatment is initiated and when dosage is changed. Capsules for each day are stored in well-marked, daily blister packs that ensure the participants are taking the correct capsules.

Treatment adherence is using weekly surveys. All botanicals used in this study are commercially available, and there are no critical reagents to obtain. The botanicals are provided by Pure Encapsulations and Nature's Way. Weekly symptom reports begin during baseline. Participants are not aware of when they change conditions, as the appearance and number of capsules are kept the same throughout participation. Symptom severity reports are provided at the end of each week for the entire duration of participation, and primary outcome assessments (the Veterans Rand 12-Item Health Survey) are also given once per week.

ELIGIBILITY:
In accordance with the Institute of Medicine (IOM) 2014 guidance, participants must meet both the Kansas and CDC (Centers for Disease Control and Prevention) Case Definitions of GWI. Participants must have been deployed to the Persian Gulf Region during the 1990-1991 Gulf War, meet symptom domain criteria, and not have exclusionary medical conditions. The case definitions will be used for inclusionary screening purposes.

Inclusion Criteria:

* Meets Kansas GWI Case Definition
* Meets CDC GWI Case Definition
* Able to commit to a 10-month study

Exclusion Criteria:

* Currently involved in an experimental treatment study
* Abnormal liver function values
* Abnormal kidney function values
* Currently pregnant
* Blood clotting disorder (contraindicated with all three botanicals)
* Reported diagnosis of diabetes with an A1C greater than 9
* The use of contraindicated medications (see below):
* Anticoagulant medications (such as warfarin, heparin, etc.)
* Lithium
* Tacrolimus (Prograf)
* Cancer medications (Alkylating agents, antitumor antibiotics, Topoisomerase I inhibitors, Tamoxifen)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Average Veterans Rand 12-Item Health Survey (VR-12) Physical Functioning Score | This outcome will be assessed weekly, for up to 44 weeks.
  Veterans Rand 12-Item Health Survey (VR-12) Physical Functioning Score (PFS) will be assessed via an online survey. The PFS will be assessed on a 7-32 point scale, with higher scores indicating better health.
Average Veterans Rand 12-Item Health Survey (VR-12) Mental Functioning Score | This outcome will be assessed weekly, for up to 44 weeks.
  Veterans Rand 12-Item Health Survey (VR-12) Mental Functioning Score (MFS) will be assessed via an online survey. The MFS will be assessed on a 6-33 point scale, with higher scores indicating better health.

SECONDARY OUTCOMES:
Patient Global Impression of Change (PGIC) | This outcome will be assessed weekly, for up to 44 weeks.
  The Patient Global Impression of Change (PGIC) assesses overall quality of life improvement and is widely used in clinical trials.
Number needed to treat (NNT) | This outcome will be assessed once, through study completion, an average of 44 weeks.
  The number needed to treat (NNT) is popular in clinical trial research and indicates the expected number of responders when used in the general GWI population.

OTHER OUTCOMES:
Weekly Symptom Reports | This outcome will be assessed weekly, for up to 44 weeks.
  The tertiary outcomes cover symptoms frequently endorsed by GWI patients. The items are designed to measure severity in all six GWI symptom domains (fatigue, pain, neurologic, skin, gastrointestinal, and respiratory). They each use a 0-100 scale. The 21 items are overall GWI severity, interference with life, muscle pain, joint pain, numbness or tingling, body tremors, fatigue, depression, stress, anxiety, irritableness/anger, sleep quality, thinking and memory quality, gastrointestinal problems, headaches, physical activity, post-exertional malaise, dizziness or faintness, respiratory issues, vision problems, and skin problems.

CONTACTS AND LOCATIONS:
Overall Officials: Jarred Younger, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Donovan EK, Kekes-Szabo S, Lin JC, Massey RL, Cobb JD, Hodgin KS, Ness TJ, Hangee-Bauer C, Younger JW. A Placebo-Controlled, Pseudo-Randomized, Crossover Trial of Botanical Agents for Gulf War Illness: Curcumin (Curcuma longa), Boswellia (Boswellia serrata), and French Maritime Pine Bark (Pinus pinaster). Int J Environ Res Public Health. 2021 Mar 3;18(5):2468. doi: 10.3390/ijerph18052468. PMID 33802272
- [Background] Hodgin KS, Donovan EK, Kekes-Szabo S, Lin JC, Feick J, Massey RL, Ness TJ, Younger JW. A Placebo-Controlled, Pseudo-Randomized, Crossover Trial of Botanical Agents for Gulf War Illness: Resveratrol (Polygonum cuspidatum), Luteolin, and Fisetin (Rhus succedanea). Int J Environ Res Public Health. 2021 Mar 3;18(5):2483. doi: 10.3390/ijerph18052483. PMID 33802381
- [Background] Younger J, Donovan EK, Hodgin KS, Ness TJ. A Placebo-Controlled, Pseudo-Randomized, Crossover Trial of Botanical Agents for Gulf War Illness: Reishi Mushroom (Ganoderma lucidum), Stinging Nettle (Urtica dioica), and Epimedium (Epimedium sagittatum). Int J Environ Res Public Health. 2021 Apr 1;18(7):3671. doi: 10.3390/ijerph18073671. PMID 33915962